CLINICAL TRIAL: NCT06096584
Title: TIPS Block vs Dual Subsartorial Block for Total Knee Arthrolplasty: Double Blinded Randomized Controlled Study
Brief Title: TIPS Block vs Dual Subsartorial Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0306191
Record Dates: First submitted 2023-10-12; First posted 2023-10-24 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia, Local; Knee Arthropathy

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TIPS (Experimental): patients will receive double level subsartorial block and suprasartorial LA injection at the level of the distal FT after induction of general anesthesia (GA)
  Interventions: Procedure: Triple Injection Perisartorius block; Procedure: Femoral triangle block; Procedure: Distal adductor canal block; Procedure: Suprasartorial plane block
- Group Dual (Active Comparator): patients will receive double level subsartorial canal block after induction of GA
  Interventions: Procedure: Dual sub sartorial block; Procedure: Femoral triangle block; Procedure: Distal adductor canal block

INTERVENTIONS:
Procedure: Triple Injection Perisartorius block — Drug: Bupivacaine 0.25 % mixed with 2 mg dexamethasone.
  Patients will receive a third injection of 10 ml of 0.25 % bupivacaine superficial to the sartorius under the facia lata
  Arms: Group TIPS
Procedure: Dual sub sartorial block — Drug: Bupivacaine 0.25 % mixed with 2 mg dexamethasone
  Patients will receive a combination of femoral triangle block and distal ACB.
  Arms: Group Dual
Procedure: Femoral triangle block — Femoral triangle block will be given just (1-2 cm) proximal to the apex of the femoral tringle which is the point at which the medial border of the sartorius muscle (STM) meets the medial border of the adductor longus muscle (ALM). Ten ml of 0.25 % bupivacaine mixed with 2 mg dexamethasone will be injected just below the STM.
Procedure: Distal adductor canal block — Another 20 ml of 0.25 % bupivacaine mixed with 2 mg dexamethasone will be injected in the lower one-third of the adductor canal.
Procedure: Suprasartorial plane block — Patients will receive a third injection of 10 ml of 0.25 % bupivacaine superficial to the sartorius under the facia lata
  Arms: Group TIPS

SUMMARY:
The present study examines adding local anesthetic injection superior to the sartorius at the level of the femoral triangle to block the intermediate femoral cutaneous nerve (IFCN) which is responsible for the innervation of the anterior thigh and the proximal part of the parapatellar incision used for total knee arthroplasty (TKA). This may provide superior analgesia when added to dual subsartorial blockade in cases of total knee arthroplasty

DETAILED DESCRIPTION:
Introduction: Maximum pain control with regional analgesic techniques after total knee arthroplasty (TKA) is crucial for early rehabilitation after surgery. The ideal regional anesthetic technique should cover all the essential innervations of the knee joint involved in each surgical step without causing motor blockade.

The investigators hypothesize that local anesthetic injection superior to the sartorius at the level of the femoral triangle may block the intermediate femoral cutaneous nerve (IFCN) which is responsible for the innervation of the anterior thigh and the proximal part of the parapatellar incision used for TKA and provide superior analgesia when added to dual subsartorial blockade in cases of TKA.

Patients will be divided into 2 groups. Group TIPS; patients will receive double level subsartorial block and suprasartorial LA injection at the level of the distal FT after induction of general anesthesia (GA). Group Dual; patients will receive double level subsartorial canal block after induction of GA.

Upon arrival to the operating room (OR), a multichannel monitor will be attached to patients, followed by the administration of 2 mg midazolam IV after securing an IV cannula. Induction of anesthesia will be carried out with 2 mic/kg fentanyl, 2 mg/kg propofol and 25 mg atracurium followed by insertion of a proper size laryngeal mask airway (LMA). Patients will be randomly allocated into 2 groups by a computer generated program.

Group Dual: Patients will receive a combination of femoral triangle block and distal ACB. Femoral triangle block will be given just 1-2 cm proximal to the apex of the femoral tringle which is the point at which the medial border of the sartorius muscle (STM) meets the medial border of the adductor longus muscle (ALM). Ten ml of 0.25 % bupivacaine mixed with 2 mg dexamethasone will be injected just below the STM. Another 20 ml of 0.25 % bupivacaine mixed with 2 mg dexamethasone will be injected in the lower one-third of the adductor canal. At this level, femoral vessels dip into the opening of the adductor hiatus to become popliteal vessels. Sonoanatomy of this region shows the adductor magnus muscle (AMM) posteromedially, vastus medialis muscle (VMM) anterolaterally, and the STM medially.

Group TIPS: Patients will receive dual injection subsartorial block and a third injection of 10 ml of 0.25 % bupivacaine superficial to the sartorius under the facia lata.

Postoperatively, multimodal analgesia regimen will be continued in the form of paracetamol 1 g /8 hours and ketorolac 30 mg /8 hours intravenously for 24 hours. Intravenous morphine patient controlled analgesia will be started after induction of GA at a concentration of 0.5 mg/ml without a background infusion on demand dose of 1 mg with a lockout interval of 10 minutes. Resting and dynamic VAS assessment will be carried out every 4 hours during the 24 hour follow up period. Total postoperative morphine requirements will be measured during the postoperative follow up period. Postoperative functional outcome will be assessed using the Timed Up and Go (TUG) test and the 30-second Chair Stand Test (30s-CST).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Scheduled for unilateral total knee arthroplasty

Exclusion Criteria:

* BMI > 35 kg/m2
* Pre-existing neurological deficit
* Any disability of the non-operated limb preventing fair mobilization
* Infection at the site of injection
* Chronic opioid users/abusers

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative resting visual analogue scale score.It's a 0-10 score where 0 is no pain and 10 is the worst pain | 1st 24 hours after surgery
  Resting visual analogue scale score assessment will be carried out every 4 hours during the 24 hour follow up period

SECONDARY OUTCOMES:
Postoperative dynamic visual analogue scale score. It's a 0-10 score where 0 is no pain and 10 is the worst pain | 1st 24 hours after surgery
  Dynamic visual analogue scale score assessment will be carried out every 4 hours during the 24 hour follow up period
Total postoperative morphine requirements | 1st 24 hours after surgery
Postoperative functional outcome | 1st 24 hours after surgery
  Timed Up and Go (TUG) test. Score < 10s indicates normal mobility
Postoperative functional outcome | 1st 24 hours after surgery
  30-second Chair Stand Test (30s-CST). The number of times the patient can stand and sit in 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analyzed during the current study are available from the corresponding author upon reasonable request
Supporting Information: Study Protocol
Time Frame: Data will be available after publication for one year
Access Criteria: moustafa.abdelaziz@alexmed.edu.eg

REFERENCES:
- [Result] Ishiguro S, Yokochi A, Yoshioka K, Asano N, Deguchi A, Iwasaki Y, Sudo A, Maruyama K. Technical communication: anatomy and clinical implications of ultrasound-guided selective femoral nerve block. Anesth Analg. 2012 Dec;115(6):1467-70. doi: 10.1213/ANE.0b013e31826af956. Epub 2012 Aug 10. PMID 22886842
- [Result] Ludwigson JL, Tillmans SD, Galgon RE, Chambers TA, Heiner JP, Schroeder KM. A Comparison of Single Shot Adductor Canal Block Versus Femoral Nerve Catheter for Total Knee Arthroplasty. J Arthroplasty. 2015 Sep;30(9 Suppl):68-71. doi: 10.1016/j.arth.2015.03.044. Epub 2015 Jun 3. PMID 26129851